CLINICAL TRIAL: NCT05488106
Title: Intervention With Riboflavin to Improve Vascular Health and ENdothelial Functioning in Genetically at- Risk Adults (InteRVENE Study)
Brief Title: Intervention With Riboflavin to Improve Vascular Health and ENdothelial Functioning in Genetically at- Risk Adults
Acronym: InteRVENE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Ulster (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC/19/0079
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Blood Pressure; Hypertension
Keywords: Blood Pressure; MTHFR; Methylenetetrahydrofolate Reductase; Riboflavin; Flow-Mediated Dilation; Nitric Oxide
MeSH Terms: conditions — Hypertension | interventions — Riboflavin

STUDY DESIGN:
Intervention Model Description: Double blind placebo controlled parallel design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Dose 1 (Active Comparator)
  Interventions: Dietary Supplement: Riboflavin 1.6mg/d
- Dose 2 (Active Comparator)
  Interventions: Dietary Supplement: Riboflavin 5mg/d
- Dose 3 (Active Comparator)
  Interventions: Dietary Supplement: Riboflavin 20mg/d

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo
  Arms: Placebo
Dietary Supplement: Riboflavin 1.6mg/d — Riboflavin 1.6mg/d
  Arms: Dose 1
Dietary Supplement: Riboflavin 5mg/d — Riboflavin 5mg/d
  Arms: Dose 2
Dietary Supplement: Riboflavin 20mg/d — Riboflavin 20mg/d
  Arms: Dose 3

SUMMARY:
High blood pressure is the leading risk factor for heart disease and stroke. Approximately 12% of the population have a particular genetic factor (known as the TT genotype) which increases the risk of high blood pressure. Previous studies conducted at this centre have shown that taking the B-vitamin riboflavin, for up to 3 months, decreases blood pressure in adults with the TT genotype. It is currently not known how riboflavin lowers blood pressure in those with the TT genotype but it could be as a result of altering blood levels of nitric oxide. Nitric oxide causes blood vessels to expand, leading to improved blood vessel function, an important predictor of cardiovascular health. However, the effect of riboflavin supplementation on nitric oxide and blood vessel function has not been previously studied. Furthermore, it is unclear whether taking riboflavin over a shorter period of time or at doses higher than 1.6 mg/d can also lower blood pressure and improve blood vessel function in this at risk group. Therefore, the aim of this study is to assess the effects of riboflavin supplementation on blood pressure, biomarkers of nitric oxide bioavailability and blood vessel function. It is hypothesised that riboflavin supplementation will increase nitric oxide bioavailability, leading to reduced blood pressure and improved blood vessel function and, and that a higher riboflavin dose will lead to greater reductions in blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 60 years and below
* Pre-screened for MTHFR 677TT genotype (TTs and CCs individuals only invited)

Exclusion Criteria:

* Consumer of B-vitamin supplements
* Consuming medication that interferes with B-vitamin metabolism

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male only
Enrollment: 120 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | Change over 16 weeks
  Branchial blood pressure
Diastolic blood pressure | Change over 16 weeks
  Branchial blood pressure

SECONDARY OUTCOMES:
Endothelial function | Change over 16 weeks
  Measured by Flow Mediated Dilation
Nitric oxide bioavailability | Change over 16 weeks
  Plasma nitrite and nitrate oxide analysed by a Sievers gas-phase chemiluminescence nitric oxide analyser
Erythrocyte glutathione reductase activation coefficient (EGRac)(Vitamin B2 marker) | Change over 16 weeks
  Measured on automatic analyser
Pyridoxal phosphate (Vitamin B6 marker) | Change over 16 weeks
  Measured on HPLC

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Ulster University, Coleraine, Co.Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Company funded work, no plan to share IPD